CLINICAL TRIAL: NCT01175018
Title: Anakinra to Prevent Adverse Post-infarction Remodeling (2)
Acronym: VCU-ART2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHA 10SDG3030051
Record Dates: First submitted 2010-07-30; First posted 2010-08-04 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Acute Myocardial Infarction; Heart Failure
Keywords: Acute myocardial infarction; Heart Failure; Cardiac Remodeling
MeSH Terms: conditions — Heart Failure | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Experimental): Anakinra 100 mg injectable subcutaneously daily
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): 0.67 ml of sodium chloride (NaCl) 0.9% solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — Anakinra 100 mg s.c. daily for 14 days
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebo — 0.67 ml of NaCl 0.9% solution given subcutaneously daily for 14 days
  Other Names: NaCl 0.9%
  Arms: Placebo

SUMMARY:
Acute myocardial infarction (AMI) remains a major cause of morbidity and mortality. Many patients die early during the course, and those who survive are at risk for dying late from adverse cardiac remodeling and heart failure.

The initial ischemic damage to the myocardium initiates an intense inflammatory response in promoting further cardiac dysfunction and heart failure. The investigators propose that an antiinflammatory strategy based on blockade of Interleukin-1 will quench the inflammatory response and lead to a more favorable cardiac remodeling process.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) remains a major cause of morbidity and mortality. Many patients die early during the course, and those who survive are at risk for dying late from adverse cardiac remodeling and heart failure.

The initial ischemic damage to the myocardium initiates an intense inflammatory response in promoting further cardiac dysfunction and heart failure. Interleukin-1 (IL-1) is the prototypical inflammatory cytokine involved in the tissue response to injury. In the experimental model of large anterior wall AMI in the mouse, IL-1 blockade using anakinra, a recombinant human IL-1 receptor antagonist ameliorates cardiac remodeling and improves survival following AMI. Although the mouse AMI model is helpful in understanding the events leading to adverse post-infarction cardiac remodeling and heart failure, the exact role of IL-1 in patients with AMI has not been completely characterized. The investigators propose to address this question by studying patients presenting with ST-segment elevation AMI (STEMI). Such patients are at high risk for in-hospital and long-term mortality and display several markers of inflammation. The investigators hypothesize that IL-1 blockade in patients STEMI with will limit the acute inflammatory response and prevent adverse cardiac remodeling, heart failure, and related morbidity.

The investigators hypothesize that treatment with anakinra will lead to more favorable cardiac remodeling. Left ventricular end-systolic volume index (LVESVi) is the preferred clinical marker of adverse cardiac remodeling and a strong predictor of heart failure-related mortality in patients with STEMI, and will be used as primary endpoint of the study. The investigators propose that anakinra will reduce the change in LVESVi from baseline to 10-14 weeks after STEMI, and will prevent, at least in part, other changes in cardiac function and exercise tolerance associated with adverse cardiac remodeling and heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI will be asked to enroll according to the following inclusion criteria:

  * age > 18 years,
  * acute (<12 h) onset of chest pain associated with ST segment elevation (>2 mm) in 2 or more anatomically contiguous leads at ECG,
  * and successful primary percutaneous coronary intervention.

Exclusion criteria:

* inability to give informed consent,
* late presentation (>12 h),
* unsuccessful revascularization procedure,
* hemodynamic instability including hypotension,
* prior Q-wave AMI,
* end-stage congestive heart failure (American Heart Association [AHA]/American College of Cardiology [ACC] class C-D, New York Heart Association IV), severe left ventricular dysfunction (EF<20%),
* severe valvular heart disease,
* pregnancy, dye allergy or contraindications to cardiac angiography and/or magnetic resonance imaging, coagulopathy (INR>1.5 or platelet count<50000/mm3),
* recent (<14 days) use of anti-inflammatory drugs (not including NSAIDs),
* chronic inflammatory disease (including but not limited to rheumatoid arthritis, systemic lupus erythematosus), and malignancy or any comorbidity limiting survival or conditions predicting inability to complete the study.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, M.D., Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbate A, Kontos MC, Grizzard JD, Biondi-Zoccai GG, Van Tassell BW, Robati R, Roach LM, Arena RA, Roberts CS, Varma A, Gelwix CC, Salloum FN, Hastillo A, Dinarello CA, Vetrovec GW; VCU-ART Investigators. Interleukin-1 blockade with anakinra to prevent adverse cardiac remodeling after acute myocardial infarction (Virginia Commonwealth University Anakinra Remodeling Trial [VCU-ART] Pilot study). Am J Cardiol. 2010 May 15;105(10):1371-1377.e1. doi: 10.1016/j.amjcard.2009.12.059. Epub 2010 Apr 2. PMID 20451681
- [Result] Abbate A, Van Tassell BW, Biondi-Zoccai G, Kontos MC, Grizzard JD, Spillman DW, Oddi C, Roberts CS, Melchior RD, Mueller GH, Abouzaki NA, Rengel LR, Varma A, Gambill ML, Falcao RA, Voelkel NF, Dinarello CA, Vetrovec GW. Effects of interleukin-1 blockade with anakinra on adverse cardiac remodeling and heart failure after acute myocardial infarction [from the Virginia Commonwealth University-Anakinra Remodeling Trial (2) (VCU-ART2) pilot study]. Am J Cardiol. 2013 May 15;111(10):1394-400. doi: 10.1016/j.amjcard.2013.01.287. Epub 2013 Feb 27. PMID 23453459
- [Derived] Abbate A, Kontos MC, Abouzaki NA, Melchior RD, Thomas C, Van Tassell BW, Oddi C, Carbone S, Trankle CR, Roberts CS, Mueller GH, Gambill ML, Christopher S, Markley R, Vetrovec GW, Dinarello CA, Biondi-Zoccai G. Comparative safety of interleukin-1 blockade with anakinra in patients with ST-segment elevation acute myocardial infarction (from the VCU-ART and VCU-ART2 pilot studies). Am J Cardiol. 2015 Feb 1;115(3):288-92. doi: 10.1016/j.amjcard.2014.11.003. Epub 2014 Nov 13. PMID 25482680
- [Derived] Sonnino C, Christopher S, Oddi C, Toldo S, Falcao RA, Melchior RD, Mueller GH, Abouzaki NA, Varma A, Gambill ML, Van Tassell BW, Dinarello CA, Abbate A. Leukocyte activity in patients with ST-segment elevation acute myocardial infarction treated with anakinra. Mol Med. 2014 Nov 18;20(1):486-9. doi: 10.2119/molmed.2014.00121. PMID 25121719
- [Derived] Falcao RA, Christopher S, Oddi C, Reznikov L, Grizzard JD, Abouzaki NA, Varma A, Van Tassell BW, Dinarello CA, Abbate A. Interleukin-10 in patients with ST-segment elevation myocardial infarction. Int J Cardiol. 2014 Mar 1;172(1):e6-8. doi: 10.1016/j.ijcard.2013.12.126. Epub 2014 Jan 5. No abstract available. PMID 24467979
- See also: VCU Pauley Heart Center — http://www.pauleyheart.vcu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra | Placebo
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1
Not completed — Adverse Event | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 0.67 ml of NaCl 0.9% solution
- Total: Total of all reporting groups
Arm/Group | Anakinra | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 58 (12) | 59 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the Anakinra Arm and the Placebo Arm in Change in Left Ventricular End-systolic Volume Indices
Description: Change in n left ventricular end-systolic volume indices from baseline to follow up exam at cardiac magnetic resonance imaging comparing anakinra- and placebo-treated patients.
Time Frame: 10-14 weeks minus baseline
Population: Applies only to subset of patients with magnetic resonance imaging (MRI) at baseline and 10-14 weeks.
Measure: Median (Inter-Quartile Range); unit: mL/m2
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
mL/m2 | 1.5 [-3 to 3] | 1.0 [-4.5 to 6]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Difference Between the Anakinra Arm and the Placebo Arm in Change in Left Ventricular End-diastolic Volume Indices From Baseline to Follow up Exam at Cardiac Magnetic Resonance Imaging
Time Frame: 10-14 weeks
Population: Applies only to subset of patients with magnetic resonance imaging (MRI) at baseline and 10-14 weeks.
Measure: Median (Inter-Quartile Range); unit: mL/m2
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
mL/m2 | 3 [-3 to 10] | -4 [-12 to 17]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

3. Secondary Outcome: Percentage of Patients in Each Group With Reverse Remodeling (Reduction in LVESVi >5%)
Time Frame: 10-14 weeks
Measure: Number; unit: % of participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
% of participants | 45 | 43
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

4. Secondary Outcome: Median Difference Between the 2 Arms in the Peak Oxygen Consumption (VO2) at 10-14 Weeks
Time Frame: 10-14 weeks
Measure: Median (Inter-Quartile Range); unit: ml*kg^-1*min^-1
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 4 | 6
ml*kg^-1*min^-1 | -1 [-13 to 1] | 2.5 [-1 to 7]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

5. Secondary Outcome: Incidence of Heart Failure
Description: Difference between the anakinra arm and the placebo arm in number of patients with a new diagnosis or admission to the hospital for heart failure
Time Frame: 10-14 weeks
Measure: Number; unit: participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 15 | 15
participants | 1 | 4
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p < 0.05, Log Rank

6. Secondary Outcome: Number of Adverse Events in Each Group
Time Frame: 10-14 weeks
Measure: Number; unit: adverse events
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 15 | 15
adverse events | 11 | 20
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

7. Secondary Outcome: Difference Between the 2 Arm in the Interval Change in Right Ventricular Ejection Fraction (RVEF)
Time Frame: 10-14 weeks
Measure: Median (Inter-Quartile Range); unit: % (absolute change)
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
% (absolute change) | 5 [-2 to 11] | 4 [-4 to 10]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

8. Secondary Outcome: Difference Between the Anakinra Arm and the Placebo Arm in Change in Left Ventricular Ejection Fraction Values From Baseline to Follow up Exam at Cardiac Magnetic Resonance Imaging
Time Frame: 10-14 weeks
Measure: Median (Inter-Quartile Range); unit: % (absolute change)
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
% (absolute change) | 2 [-2 to 10] | -2 [-5 to 5]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

9. Secondary Outcome: Median Difference Between the 2 Arms in the Ratio of Minute Ventilation and Carbon Dioxide Production (VE/VCO2 Slope) at 10-14 Weeks
Time Frame: 10-14 weeks
Measure: Median (Inter-Quartile Range); unit: (no units; ratio of values)
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 4 | 6
(no units; ratio of values) | -1 [-17 to 2] | -3 [-6 to -1]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

10. Secondary Outcome: Percentage of Patients in Each Group With Reverse Remodeling (Reduction in LVESVi >10%)
Time Frame: 10-14 weeks
Measure: Number; unit: % of participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
% of participants | 27 | 36
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

11. Secondary Outcome: Percentage of Patients in Each Group With Adverse Remodeling (LVESVi Increase >5%) Based Upon Cardiac Magnetic Resonance Imaging
Time Frame: 10-14 weeks
Population: Applies only to subset of patients with magnetic resonance imaging (MRI) at baseline and 10-14 weeks.
Measure: Number; unit: % of participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
% of participants | 55 | 42
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

12. Secondary Outcome: Percentage of Patients in Each Group With Adverse Remodeling (LVESVi Increase >10%)
Time Frame: 10-14 weeks
Measure: Number; unit: % of participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
% of participants | 45 | 29
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

13. Secondary Outcome: Percentage of Patients in Each Group With Left Ventricular Ejection Fraction Change >5%
Time Frame: 10-14 weeks
Measure: Number; unit: % of participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
% of participants | 36 | 36
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

14. Secondary Outcome: Percentage of Patients in Each Group With Left Ventricular Ejection Fraction Change >10%
Time Frame: 10-14 weeks
Measure: Number; unit: % of participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 11 | 14
% of participants | 27 | 0
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

15. Secondary Outcome: Number of Deaths in Each Group
Time Frame: 10-14 weeks
Measure: Number; unit: deaths
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 15 | 15
deaths | 0 | 1
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

16. Secondary Outcome: Number of Adverse Events Requiring Withdrawal in Each Group
Time Frame: 10-14 weeks
Measure: Number; unit: adverse events
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 15 | 15
adverse events | 2 | 2
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Anakinra | Placebo
Serious Adverse Events (participants affected / at risk) | 4/15 | 6/15
Other Adverse Events (participants affected / at risk) | 6/15 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=15) | Placebo (N=15)
Death (Cardiac disorders) | 0 (0) | 1 (1)
New onset heart failure (Cardiac disorders) | 1 (1) | 4 (4)
Serious infection (Infections and infestations) | 2 (2) | 2 (2) — requiring or prolonging hospital admission, or requiring intravenous antibiotics
Recurrent myocardial infarction or repeat percutaneous coronary intervention (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac rupture (Cardiac disorders) | 0 (0) | 1 (1) — Cardiac rupture
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=15) | Placebo (N=15)
Bleeding (not serious) (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Injection site pain (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection (not serious) (Infections and infestations) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes